CLINICAL TRIAL: NCT05859828
Title: A sinGle-arm Phase 2 Study to Assess Efficacy, tOxicity, and quAlity of Life Following 27Gy in 6 Fractions Palliative Intensity Modulated Radiotherapy in Advanced Head and Neck Cancer
Brief Title: The GOAL27-6 Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: East and North Hertfordshire NHS Trust (Other Government)
Collaborators: Get A-Head Charitable Trust (Unknown)
Responsible Party: Sponsor
Other Study IDs: RD2021-44
Record Dates: First submitted 2023-05-05; First posted 2023-05-16 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Head and Neck Cancer patients: Participants with incurable advanced head and neck cancer. Participants will have histologically or cytologically confirmed squamous cell carcinoma of the head and neck
- Patient Caregivers: Caregivers to participants in the patient cohort

SUMMARY:
The main purpose and goal of this study is to find out if a particular course of radiotherapy for non-curable cancers, together with palliative care support, can help improve patients' quality of life.

DETAILED DESCRIPTION:
Approximately a quarter of head and neck cancer patients are unfortunately not deemed curable. This is either due to the late advanced nature of the cancer at presentation, or patient's limited medical fitness to go through the intensive curative treatment. With the incurable growing cancer, these patients commonly have debilitating symptoms such as pain, discharge or bleeding that could adversely affect their quality of life and that of their caregivers. As well as palliative care input, palliative radiotherapy is given with the aim of relieving these symptoms.

There is a wide variation in the palliative radiotherapy practice locally and internationally. Despite the differences, the paradigm certainly is that higher dose radiotherapy does not necessarily mean better palliation, as high dose radiation itself could lead to more treatment toxicity, which could affect the quality of patients' limited life expectancy.

Intensity modulated radiotherapy (IMRT) is a more precise treatment known to offer fewer toxicity than the traditional (non-IMRT) radiotherapy. Not all centres in the UK offer palliative head and neck radiotherapy using IMRT. As a high volume centre, Mount Vernon has the experience of delivering palliative head and neck IMRT almost as quick as the non-IMRT technique. One of the departmental palliative regimens is 27Gy in 6 fractions, with treatment twice a week for 3 weeks.

Since the implementation of IMRT with for this dose fractionation in 2019, there has been noticeable improvement in patients' quality of life as well as their caregivers. This is however anecdotal, and the aim of this study is to objectively evaluate this practice using validated quality of life questionnaires

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and over
* Histologically or cytologically confirmed squamous cell carcinoma of the head and neck
* Neck disease from cutaneous squamous cell carcinoma of head and neck area
* Measurable disease on clinical examination (e.g. transoral examination, neck palpation) for post-radiotherapy comparison or if no assessable disease at baseline, patient will have disease amenable to post-radiotherapy investigations of response per SOC
* Patients not clinically deemed to be suitable for radical / curative surgery or radiotherapy
* Life expectancy of at least 3 months
* Patient due to undergo 27Gy in 6f palliative radiotherapy outside the study
* Capable of providing written or witnessed informed consent according to ICH/GCP and national/local guidelines prior to registration
* Patients consent to hospital and/or community palliative care referrals

Inclusion Criteria for carers

* consent is needed from the patient for carer involvement
* carers should have adequate command of English language to read and answer questionnaires
* capable of at least providing written or witnessed informed consent

Exclusion Criteria:

* Non squamous cell carcinoma of the head and neck
* Previous radiotherapy to the head and neck
* Palliative systemic treatment (chemotherapy/immunotherapy) given prior to palliative radiotherapy. Subsequent systemic treatment is allowed on progression of disease after palliative radiotherapy.
* ECOG performance status 4
* Any psychological, familial, sociological or geographical condition in patients or carers potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the participant before registration in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Head and neck squamous cell cancer patients, where palliative radiotherapy is the treatment. Up to 30 carers will also be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-04-21 (Actual); Primary Completion 2024-04-21 (Estimated); Study Completion 2025-04-21 (Estimated)

PRIMARY OUTCOMES:
Patient quality of life (QoL) in head and neck cancer patients receiving 27 Gray (Gy) in 6 fractions (f) palliative Intensity Modulated Radiotherapy (IMRT). | 12 months
  measured via scores on validated FACT-HN questionnaire
Toxicity (Grade 3 or worse) in head and neck cancer patients receiving 27 Gray (Gy) in 6 fractions (f) palliative Intensity Modulated Radiotherapy (IMRT). | 12 months
  measurement as per Common Terminology Criteria of Adverse Events v5.0

SECONDARY OUTCOMES:
Caregiver quality of life following patients receiving 27Gy in 6f IMRT | 12 months
  Assessed via the CarGoQol questionnaire

OTHER OUTCOMES:
Patient survival following 27 Gray (Gy) in 6 fractions (f) palliative Intensity Modulated Radiotherapy (IMRT). | 12 months
  Measured by Overall Survival (OS) and Progression Free Survival (PFS)
Patient response following 27 Gray (Gy) in 6 fractions (f) palliative Intensity Modulated Radiotherapy (IMRT). | 12 months
  Classified as either Complete response, Partial Response, stable disease or progressive disease

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Vernon Cancer Centre, Northwood, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
The research results will be published in international journals and presented at scientific meetings.